CLINICAL TRIAL: NCT02109497
Title: A Phase 1, Single Centre, Open Label, Two-period Study in Healthy Volunteers to Determine the Effect of PBT2 on the Pharmacokinetics of Caffeine
Brief Title: Phase 1 Study to Determine the Effects of PBT2 on the Pharmacokinetic Profile of Caffeine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prana Biotechnology Limited (Industry)
Responsible Party: Sponsor
Organization: Pranabio (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBT2-104
Record Dates: First submitted 2014-04-03; First posted 2014-04-10 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caffeine Dosing (Other): Single dose of caffeine 100 mg administered
  Interventions: Drug: PBT2

INTERVENTIONS:
Drug: PBT2 — PBT2 250 mg administered

SUMMARY:
This study is designed to determine the pharmacokinetic (PK) profile of a single oral dose of caffeine and the effects that PBT2 has on the metabolism of caffeine in healthy volunteers.

DETAILED DESCRIPTION:
This study will be conducted with all participants receiving a dose of caffeine 100 mg on Day 1 followed by a 7 day washout period before commencing 5 consecutive days of PBT2 250 mg from Day 8 to 12 and a second dose of caffeine 100 mg on Day 12. Pharmacokinetic samples will be collected during after each dose of the study drugs, along with safety monitoring assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females with a BMI between 19 and 30kg/m2
* No clinically significant abnormalities

Exclusion Criteria:

* Exposure to medications/drugs that interfere with metabolism of PBT2 including drugs that inhibit or induce CYP1A2
* Use of caffeine-containing beverages, supplements or alcohol
* Significant history of depression or other psychiatric illness
* Surgical or medical conditions which could significantly alter drug absorption, distribution, metabolism or excretion
* Unable to swallow capsules or tablets

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Herd, Study Director — Prana Biotechnology
Locations (1):
- Centre for Clinical Studies - Nucleus Network, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled at one study site in Australia
Groups:
- Caffeine Dosing: Single dose of caffeine 100 mg administered on Day 1 and Day 12 with PBT2 250 mg administered from Day 8 to 12.
Period: Overall Study
Arm/Group | Caffeine Dosing
Started | 18
Completed | 17 (One participant completed the safety assessments but did not complete all doses of the study drugs.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Caffeine Dosing: Single dose of caffeine 100 mg administered on Day 1 and Day 12
  PBT2: PBT2 250 mg administered is Day 8 to 12.
Arm/Group | Caffeine Dosing
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Australia | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.05 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Caffeine After a Dose of PBT2 250mg
Description: PK Per Protocol Population, as defined as all participants who received scheduled doses of both caffeine and PBT2 and had sufficient samples collected to determine PK parameters from plasma concentrations of caffeine on Day 1 and Day 12.
Time Frame: prior to dose on Day 1 and 12 and then 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 30, 36, 48 hours post each dose.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Caffeine Dosing
Number analyzed (Participants) | 17
ng*hr/mL | 32775 (11552)

2. Secondary Outcome: Safety and Tolerability of PBT2 in Healthy Volunteers Measured by the Number of Participants Reporting at Least One Treatment Emergent Adverse Event
Time Frame: Up to 19 days after first dose of caffeine
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Caffeine Dosing
Number analyzed (Participants) | 18
participants | 7

ADVERSE EVENTS:
Time Frame: All adverse events reported from time of consent to end of study (Day 19, which was 7 days since last dose of both caffeine and PBT2).
Arm/Group | Caffeine Dosing
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 7/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caffeine Dosing (N=18)
Nausea (Gastrointestinal disorders) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less